CLINICAL TRIAL: NCT02386007
Title: A Double-blind, Multicenter, Randomized Phase 2a Study to Evaluate Optimum Dosage and Stability of DW-3101 in Korean Patients With Gastric Inflammation
Brief Title: Phase 2a Study to Evaluate Optimum Dosage and Stability of DW-3101 in Gastric Inflammation Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW 3101_201
Record Dates: First submitted 2015-02-16; First posted 2015-03-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Acute and Chronic Gastric Inflammation Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- DW-3101_150mg (Experimental): 150mg a day
  Interventions: Drug: DW-3101_150mg
- DW-3101_300mg (Experimental): 300mg a day
  Interventions: Drug: DW-3101_300mg
- DW-3101_600mg (Experimental): 600mg a day
  Interventions: Drug: DW-3101_600mg
- a tablet same as experimental agents in formation and shape (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DW-3101_150mg
  Arms: DW-3101_150mg
Drug: DW-3101_300mg
  Arms: DW-3101_300mg
Drug: DW-3101_600mg
  Arms: DW-3101_600mg
Drug: Placebo
  Arms: a tablet same as experimental agents in formation and shape

SUMMARY:
The purpose of this study is to find optimum dosage of DW-3101 by evaluating efficacy and safety of each dosage group in Korean patients with acute and chronic gastric inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adult males/females aged 20~75 years
* Patients detected over 1 erosion who diagnosed as acute or chronic gastric inflammation by gastrscopy in 7days before administration of experimental agents
* Subjects who voluntarily agree to participate in this clinical test with written consent

Exclusion Criteria:

* Patients impossible gastroscopy
* In case accompanied with gastric ulcer(scar excepted) or reflux esophagitis
* Patients who had stomach or esophagus surgery to inhibit gastric acid secretion (tresis or appendicectomy surgery excluded)
* Patients with malignant tumor on digestive organ
* Patients with blood clot(cerebral thrombosis, myocardial infarction, septic thrombophlebitis) and who have antithrombotic agents (eg. warfarin)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The change of gastric erosion score | 14day±3
  The erosion score is evaluated by gastroscopy. Erosion score The number of erosion
  1. 0
  2. 1~2
  3. 3~5
  4. More than 6 If patient's erosion score is decreased by 50% compared with erosion score before clinical dosing, we count it as effectiveness.